CLINICAL TRIAL: NCT03112993
Title: A Prospective, Randomized, Double-Blind Clinical Trial Evaluating the Speed of Recovery and Safety of Reversal of Neuromuscular Blockade With Sugammadex (Bridion™) Versus Neostigmine in Geriatric Patients Undergoing Spine Surgery
Brief Title: Speed of Recovery of Reversal of Neuromuscular Blockade in Geriatric Patients Undergoing Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Boris Mraovic, Professor of Clinical Anesthesiology, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB # 2008066; MISP # 56051. (Other Grant/Funding Number: Merck & Co.)
Record Dates: First submitted 2017-03-29; First posted 2017-04-13 (Actual); Results first posted 2020-02-10 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Spine Surgery
Keywords: spine surgery; neuromuscular blockade; sugammadex; elderly; reversal; neostigmine; recovery
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Intervention Model Description: Participants will receive (per a randomization schedule) either sugammadex, or neostigmine/glycopyrrolate to reverse neuromuscular blockade at the end of the surgery. The reversal agent will be prepared in a blinded fashion.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The surgeon, anesthesiologist, operating room staff, patients, personnel in the postanesthesia care unit (PACU) as well as the investigators collecting the postoperative data will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sugammadex group (Experimental): 2 mg/kg of sugammadex, IV once at the end of the surgery. Dosing will be based on actual body weight not ideal body weight.
  Interventions: Drug: sugammadex
- Neostigmine group (Active Comparator): 50 micrograms/kg (not to exceed 5 mg) and glycopyrrolate, 10 micrograms/kg (not to exceed 1 mg), IV once at the end of the surgery.
  Dosing will be based on actual body weight not ideal body weight.
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: sugammadex — once at the end of the surgery
  Other Names: Bridion
  Arms: Sugammadex group
Drug: Neostigmine — once at the end of the surgery
  Arms: Neostigmine group

SUMMARY:
Spine surgery is one of the most common operative procedures in the United States. It is performed in the prone position (a patient laying on belly). Muscle relaxants are given for neuromuscular blockade often referred as paralysis for surgical exposure which is maintained until the patient is returned to the supine position (a patient laying on back) at the end of surgery. At the end of the surgery the paralysis is reversed with a drug (neostigmine). A new drug (sugammadex) has the ability to rapidly reverse the paralysis but it is not well investigated in elderly. This study will investigate speed of recovery and complications of the two reversal drugs in elderly patients (age ≥ 65 years) undergoing posterior spine surgery.

DETAILED DESCRIPTION:
The elderly (age ≥ 65 years) population is the fastest growing segment of the American population. Spine surgery is one of the most common operative procedures in the United States and, as the population ages, a larger percentage of geriatric patients will require this procedure. In addition, spinal surgery is often more complex in the elderly population, resulting in longer surgical times. A previous study reported that the rate of complex procedures increased 15-fold in Medicare recipients. Spine surgery is performed in the prone position and neuromuscular blockade (NMB) is maintained until the patient is returned to the supine position at the end of surgery to avoid the risk of patient movement, injury, and inadvertent tracheal extubation while prone. Currently, NMB is reversed with neostigmine immediately after turning the patients back to the supine position at the end of the procedure.

Rocuronium bromide, an intermediate-acting neuromuscular blocking agent (NMBA), is used in approximately 60% of surgical cases in the United States and is commonly used for muscle relaxation during spinal surgery. With aging, the clearance and half-life of rocuronium is prolonged resulting in a wide variability in the duration of action and time to reversal. Until recently, the only medication available for the reversal of neuromuscular blockade was neostigmine and postoperative residual neuromuscular block (PRNB) was common, especially in elderly patients. A recent study reported that PRNB occurred in 58% of elderly patients who were maintained at a moderate level (2 twitches in the TOF) of muscle relaxation with rocuronium during elective surgery. As a result, these older adults experienced an increased incidence of airway obstruction, hypoxemic events, muscle weakness, postoperative pulmonary complications, and increased PACU and hospital lengths of stay.

A new neuromuscular reversal agent sugammadex (Bridion®) has the ability to rapidly reverse both moderate and deep rocuronium-induced NMB. Another study reported that the mean time to complete reversal (TOF ratio ≥ 0.9) of a moderate block (2 twitches in the TOF) with sugammadex in geriatric patients was 2.9 minutes, which was only 1 minute longer than in younger patients. Reversal of NMB with neostigmine is much slower and it is reported to take approximately 19 minutes to achieve complete reversal in middle-aged patients. There is little available data on the NMB reversal time in older adults, but it will likely be even longer because the age-related physiologic changes prolong neuromuscular recovery. Thus, sugammadex has the potential to more rapidly reverse NMB in geriatric patients at the end of surgery. As a result, the use of sugammadex should decrease time in the OR and possibly PACU time and result in cost savings.

Neostigmine has cardiac muscarinic effects and, therefore, has to be administered with an anticholinergic agent such as glycopyrrolate to counteract these effects. A previous study found a 16% incidence of cardiac dysrhythmias in elderly patients who received neostigmine/glycopyrrolate NMB reversal. The ability of sugammadex to completely reverse NMB without the addition of an anticholinesterase agent should result in an improved safety profile in elderly patients.

The goal of this prospective, randomized, double-blinded controlled trial is to test the hypothesis that the reversal of neuromuscular blockage with sugammadex as compared to neostigmine in geriatric patients will provide a shorter time to complete recovery of neuromuscular function, improve the workflow in the operating room and decrease operative costs.

ELIGIBILITY:
Inclusion Criteria:

1. Posterior spinal surgery
2. Age ≥ 65 years
3. American Society of Anesthesiologists (ASA) grade I-III

Exclusion Criteria:

1. Inability to obtain written informed consent
2. Allergy to rocuronium or anesthetic agents used in the protocol
3. Known or suspected neuromuscular disorders
4. Significant renal disease with a serum creatinine ≥ 2 mg/dl
5. Significant liver disease
6. A family history of malignant hyperthermia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Mraovic, MD, Principal Investigator — Univesity of Missouri-Columbia
Locations (1):
- University on Missouri Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mraovic B, Timko NJ, Choma TJ. Comparison of recovery after sugammadex or neostigmine reversal of rocuronium in geriatric patients undergoing spine surgery: a randomized controlled trial. Croat Med J. 2021 Dec 31;62(6):606-613. doi: 10.3325/cmj.2021.62.606. PMID 34981693

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period
  First subject on study: 30/MAY/2017; Last subject off study: 14/AUG/2018.
  Locations: University Hospital and Missouri Orthopaedic Institute, University of Missouri, Columbia, Missouri, United States of America.
Groups:
- Neostigmine Group: 50 micrograms/kg (not to exceed 5 mg) and glycopyrrolate, 10 micrograms/kg (not to exceed 1 mg), IV once at the end of the surgery.
  Dosing will be based on actual body weight not ideal body weight.
  Neostigmine: once at the end of the surgery
Period: Overall Study
Arm/Group | Sugammadex Group | Neostigmine Group
Started | 19 | 21
Completed | 19 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex Group | Neostigmine Group | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (4.7) | 71.2 (4.8) | 70.8 (4.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 10 | 17 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 18 | 20 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ASA Physical Status Classification [Count of Participants; unit: Participants] — American Society of Anesthesiologists (ASA) physical status (PS) classification system (scale range: ASA PS 1-6). Per study protocol, subject inclusion was dependent on classification as ASA PS 1-3 and these groups can be described as follows: ASA PS 1 (a normal healthy patient); ASA PS 2 (a patient with mild systemic disease); ASA PS 3 (a patient with severe systemic disease). ASA PS classification is determined by the anesthesiologist on the day of surgery following subject interview and physical assessment.
  Participants
    ASA PS 2 | 8 | 5 | 13
    ASA PS 3 | 11 | 16 | 27
Duration of surgery [Mean (Standard Deviation); unit: minutes] | 175 (128) | 196 (96) | 185.5 (112)
End of surgery to administration of reversal (min) [Mean (Standard Deviation); unit: minutes] | 5.5 (2.0) | 4.8 (1.4) | 5.15 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Time of Neuromuscular Recovery From a Neuromuscular Moderate Blockade
Description: Speed of neuromuscular recovery in minutes measured by recovery of the T4:T1 ratio ≥ 0.9 (measured with a TOF-Watch SX)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Sugammadex Group: 2 mg/kg of sugammadex, IV once at the end of the surgery.
  Dosing will be based on actual body weight not ideal body weight.
  sugammadex: once at the end of the surgery
Arm/Group | Sugammadex Group | Neostigmine Group
Number analyzed (Participants) | 19 | 21
Minutes | 3.9 (2.2) | 26.29 (17.51)

2. Primary Outcome: Difference in Time From Neuromuscular Reversal to Exit From OR
Description: Difference in time from neuromuscular reversal to exit from OR was measured in minutes.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex Group | Neostigmine Group
Number analyzed (Participants) | 19 | 21
minutes | 3.9 (2.2) | 19.8 (13.8)

3. Secondary Outcome: Difference in Time From Neuromuscular Reversal to Tracheal Extubation
Description: Difference in time from neuromuscular reversal to tracheal extubation was measured in minutes.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex Group | Neostigmine Group
Number analyzed (Participants) | 19 | 21
minutes | 5.3 (2.5) | 23.6 (18.7)

4. Secondary Outcome: Difference in Length of Stay in PACU
Description: Length of PACU stay measured in minutes.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sugammadex Group | Neostigmine Group
Number analyzed (Participants) | 19 | 21
minutes | 81.4 (16.5) | 85.3 (29.5)

5. Other Pre Specified Outcome: Difference in Time to First Ambulation After Surgery
Description: Time from end of anesthesia to the first subject ambulation in hours.
Time Frame: From Day 1 up to 1 week, depending on individual recovery time
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sugammadex Group | Neostigmine Group
Number analyzed (Participants) | 19 | 21
hours | 17.4 (14.6) | 17.8 (11.1)

ADVERSE EVENTS:
Time Frame: Each subjects was assessed for all-cause mortality, serious adverse events, and other adverse events across their entire duration of study participation, which was the time a subject provided written informed consent until their inpatient hospital discharge following surgery. This time frame was on average 4 days.
Description: All-cause mortality, serious adverse events, and other adverse events were systematically assessed by study physician investigators through regular investigator assessment, and through review of subjects' electronic medical records during study participation.
Arm/Group | Sugammadex Group | Neostigmine Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 2/19 | 4/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sugammadex Group (N=19) | Neostigmine Group (N=21)
ICU admission (Surgical and medical procedures) | 0 | 1 — Unanticipated ICU admission due to surgical bleeding
Blood transfusion (Surgical and medical procedures) | 1 | 2 — Perioperative blood transfusion
Prolonged hospitalization (Surgical and medical procedures) | 2 | 2 — Longer hospital stay than anticipated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT03112993/Prot_SAP_000.pdf